CLINICAL TRIAL: NCT06588062
Title: Effect of Picture Exchange Communication System in Improving Oral Hygiene Status Among Preschool Children with Autism Spectrum Disorder-A Randomized Controlled Trial
Brief Title: Effect of PECS in Improving Oral Hygiene Status Among Preschool Chidren
Acronym: PECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Saqib Minhas, MDS Trainee, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB-2823/DUHS/Approval/2022/57
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: oral health status; child; preschool; autism spectrum disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group I (Experimental): All the participants of intervention (Group I) will receive conventional oral hygiene instructions in presence of their parents. These instructions will be given on model, showing each surface to be cleaned properly. Tooth brushing with the Horizontal Scrub Technique will be promoted and performance of brushing twice daily for 2 minutes. Moreover, avoidance of sugary diet will also be given. In addition the intervention participants (Group I) will be provided with PECS tool to be utilized during tooth brushing. It will be a set of 10 picture cards depicting brushing sequence and techniques by animated character. The picture will be illustrating brushing of left and right buccal, lingual, labial, and occlusal surfaces of maxillary and mandibular teeth. Each card will be accompanied by the instructions of specific step of technique with clear picture illustration for better understanding. The same instructions will be provided again, one week apart for development of skills.
  Interventions: Other: Picture Exchange Communication System (PECS)
- Control Group II (No Intervention): All the participants of control (Group II) will receive conventional oral hygiene instructions in presence of their parents. These instructions will be given on model, showing each surface to be cleaned properly. Tooth brushing with the Horizontal Scrub Technique will be promoted and performance of brushing twice daily for 2 minutes. Moreover, avoidance of sugary diet will also be given. However, PECS tool is not used as an intervention in this group. The same instructions will be provided again, one week apart for development of skills.

INTERVENTIONS:
Other: Picture Exchange Communication System (PECS) — Picture exchange communication System (PECS) is a widely useful tool for developing skills in ASD children. Visual supports rather work better for their intellectual level as these children usually respond less to verbal and written instructions. PECS is considered as an augmentative communication system commonly used with non-verbal ASD children. It is helpful for an individual with ASD to quickly acquire a functional means of communication. This is highly beneficial for the child to communicate with his parents and caregivers, as well as with their peers. Moreover, the pictorial approach of PECS is a source of facilitating element in attaining student's concentration. The reason for wide acceptance of this tool in clinical and social settings for children with ASD is its' ease of use, ability to teach two-way communication and inexpensiveness. PECS has demonstrated successful use in teaching various skills in ASD affected children lacking speech.
  Arms: Intervention Group I

SUMMARY:
Background:

Oral health is an important part of overall health of the children and precisely it is additionally imperative for children who need out of the ordinary or special health care. Children with autism spectrum disorder normally face trouble in maintenance of good oral hygiene due to their incapacity to communicate and interact socially and are one such group lacking sufficient oral health knowledge to sustain their oral health owing to communication barriers.

Objective:

To assess and compare the effect of Picture Exchange Communication System (PECS) intervention on oral hygiene status of preschool children (aged 4 to 6 years old) with Autism Spectrum Disorder (ASD) over a period of three months.

Methods:

Children with confirmed diagnosis of autism will be randomly divided into two groups. All the participants of both the groups, intervention (Group I) and control (Group II) will receive conventional oral hygiene instructions in presence of their parents. These instructions will be given on model, showing each surface to be cleaned properly. Tooth brushing with the Horizontal Scrub Technique will be promoted and performance of brushing twice daily for 2 minutes. Moreover, instruction to avoid sugary diet will also be given. Additionally, the intervention participants (Group I) will be provided a set of 10 picture cards depicting brushing sequences and techniques by animated character for PECS intervention. The plaque scores will be recorded in the two groups by using PI index by Silness & Loe (1964), GI scores will also be recorded by using GI index Loe & Silness (1963) using a periodontal probe at baseline. Following the initial examination, oral health education will be given on model to both groups, in addition to this (Group I) will be demonstrated to use PECS intervention. After three months follow up visit will be conducted in which plaque and gingival scores will be recorded again in both groups to assess the impact of PECS intervention on oral hygiene status of children with ASD.

DETAILED DESCRIPTION:
RATIONALE OF STUDY The population with Autism Spectrum Disorder Syndrome (ASD) may require additional specific health needs due to their characteristic features. Among them especially children are at risk of many diseases due to major barriers that are found in improving health and wellbeing, because of lacking in health infrastructure in Pakistan. There is vast knowledge gap and very limited research is available on this subject specially when investigated in context of Pakistan. The scenario also worsens due to delayed diagnosis and treatment intervention to this population, whereas when it comes to dental needs major factors are responsible for its unmet treatment needs. The most important factors observed are lack of access to dental consultation, affordability and refraining treatment provision by dentist as these children are sensitive to many stimuli due to which their cooperation and management is usually compromised. This shows that it is essential to identify such existing voids and take remedial measures for it. Evidence based behavioral management approaches will be key to develop and improve compliance with oral health for patients with ASD. ASD children have difficulty in communication which leads to inability to interact socially. This is due to their altered behavior patterns which includes restricted, repetitive and stereotyped pattern of behavior. Due to behavioral issues there is lack of compliance to maintenance of oral health. As a result oral health is compromised and since the behavioral component makes them difficult to interact with the dentist, their treatment management also gets difficult. Hence focus should be done on prevention of oral diseases. PECS is an effective behavioral tool for teaching ASD children basic oral health maintenance techniques. In a low socioeconomic country like Pakistan where such disabled population is not given appropriate resources and workforce, improving oral health status of such population through a cost effective technique like PECS may help lower the burden of the disease from ASD children.

Since majority of studies have not been done as a case-control, interventional or prospective cohort, however most researches have not demonstrated or compared different technique / techniques nor mentioned the comparison in-between the technique, for instance the use of PECS with other conventional methods. Therefore, this study has been undertaken to carry out a randomized controlled trail, using blinding to keep the information and results as confidential and authentic as possible. For this reason, this research will compare PECS (test) with controls (conventional method) for providing a comparative analysis as well as provide most reliable evidence on the effectiveness of the intervention by minimizing risk of confounding factors which will influence the results.

STATEMENT OF PROBLEM Pakistan is considered as a Developing country with total population of 216.6 million as of 2019. Despite of huge population Pakistan is trying to improve different sectors in different aspects including health care delivery system. Unfortunately, the health sector framework and infrastructure is still delivering poor quality and working in inefficient manner at many different levels due to many reasons. Situation is found even worse for special population which includes people with disabilities, mental health issues, developmental and neurological disorder. Similarly, the scenario is not much differing for developmental and neurological disorder including ASD as well. This lacking is observed almost at every level of policy making and implementation. There is serious lacking in providing good institutions for their development, health, education and promotion. However, the scenario is same with oral health status and its promotion among autistic children in our country. Though the disorder is not rare but as compared to developed countries relatively little reflection and attention has been drawn towards it. Usually, the attention is not drawn because people affected with autism are subject to stigma and discrimination. As ASD children have difficulty in communication which leads to inability to interact socially due to their altered behavior patterns. Due to these communication and behavioral issues there is lack of compliance to maintenance of oral health. As a result oral health is compromised and since the behavioral component makes them difficult to interact and communicate with the dentist, their treatment management also gets difficult. Hence focus should be done on prevention of oral diseases. Picture Exchange Communication System is one widely used approach to communicate and develop skills in these children.

HYPOTHESIS:

Null Hypothesis (HO) There is no effect of Picture Exchange Communication System (PECS) on oral hygiene status of preschool children with Autism Spectrum Disorder (ASD)

Alternate Hypotheses (HA) There is effect of Picture Exchange Communication System (PECS) on oral hygiene status of preschool children with Autism Spectrum Disorder (ASD)

SAMPLING TECHNIQUE:

Purposive sampling technique will be used in this study. After application of inclusion and exclusion criteria, the selected children will be allocated in groups through randomization.

RANDOMIZATION:

Sequence Generation:

After application of inclusion and exclusion criteria the selected 80 children will be numbered in the form of a list. Each eligible child will be randomly allocated to interventional and control group via SNOSE.

Allocation Concealment:

Allocation to PECS intervention (GROUP I) and control (GROUP II) will be done by Sequentially Numbered Opaque Sealed Envelope (SNOSE). The allocation of participants in intervention and control group will be written on paper and kept in a sealed and labeled envelope with a serial number on it. The researcher will assure the participants' details before envelopes are opened.

The study will follow a single blind criterion wherein the participant and their parent/caregiver will not be informed about the enrolment into which group.

DATA COLLECTION PROCEDURE:

RECRUITMENT AND ASSESSMENT:

Parents of eligible children at organizations will be invited to participate in this clinical trial with their ASD affected child. They will be provided with informed assent and details of study. The written consent will be signed by each participant's parent. Data will be collected by administering a questionnaire inquired from parent or guardian and by performing oral examinations of the participants. Performa will consist of demographic profile and autism assessment score. The demographic profile will include information related to gender, age, ethnicity, medical history, family income and parents' education. Moreover, information about previous interaction with Picture Exchange Communication System will also be included in this part of questionnaire.

The autism assessment score will be achieved from special needs organization where the child in enrolled. ASD and its severity will be assessed on the basis of CARS (Childhood Autism Rating Scale). At all special needs organization a qualified psychologist carries out CARS assessment of ASD children prior to recruitment and administration of therapies in routine. Only children with mild to moderate CARS score in the range of 30-36.5 will be enrolled in this study. If in case severity exceeds from required criteria above 37 then subjects will be excluded from the study at baseline as mentioned in the inclusion criteria. Moreover, this score will also be helpful in assessing cooperation level during oral examination.

ORAL EXAMINATION:

BASELINE EXAMINATION:

The oral examination will be performed at baseline of each study participant. This examination will be performed by principal investigator (Dr. Saqib Minhas) by using sterilized periodontal probe (Michigan-O Probe), mouth mirrors, and explorer under artificial light source. Oral examinations will be carried out on the mobile dental unit at their respective institute. Oral hygiene status will be assessed by using plaque index (PI) whereas gingival status by using gingival index (GI). The principal researcher will be trained and calibrated for intra examiner reliability for evaluation of oral hygiene indices. For the purpose a pilot study will be conducted on 20% of total sample size. And intra examiner reliability score of more than 80% will be acceptable. Both indices' readings of each participant will be recorded in Performa according to criteria of scoring i.e. GI readings are recorded as 0.1-1 (Mild), 1.1-2 (Moderate) and 2.1-3 (Severe) while for PI 0 (Excellent), 0.1-0.9 (Good), 1-1.9 (Fair), 2-3 (Poor). The following six index teeth (Ramfjord teeth) will be utilized to record PI and GI in the primary dentition (55, 61, 64, 75, 81, 84) according to the FDI system.(24) An assistant will be available at all follow ups to assist the clinician.

INTERVENTION

All the participants of both the groups, intervention (Group I) and control (Group II) will receive conventional oral hygiene instructions in presence of their parents. These instructions will be given on model, showing each surface to be cleaned properly. Tooth brushing with the Horizontal Scrub Technique will be promoted and performance of brushing twice daily for 2 minutes. Moreover, avoidance of sugary diet will also be given. The intervention participants (Group I) will be provided a set of 10 picture cards depicting brushing sequence and techniques by animated character.(24) The picture will be illustrating brushing of left and right buccal, lingual, labial, and occlusal surfaces of maxillary and mandibular teeth. The same systematic brushing steps and cleaning of all teeth and their surfaces will be demonstrated to their parents as well. However, PECS tool is used as is to avoid modification to the source. (24) Each card will be accompanied by the instructions of specific step of technique with clear picture illustration for better understanding. The same instructions will be provided again, one week apart for development of skills.

Final follow-up appointment will be scheduled at an interval of three months after intervention is applied. If in case parents and child are unable to attend appointment, reschedule will be done. Three attempts will be made for rescheduling of follow-ups.

FOLLOW UP EXAMINATION:

Follow up will be conducted after one month and two month of baseline readings where reinforcement of technique will be performed and adherence will be assessed. Oral examination will be conducted after three months in a similar manner as conducted at the time of baseline examination. The reason for selecting three month follow up is that PI can be changed over a very short period of time depending on tooth brushing (24). There are evidences that testified an oral health promotion program using both group education and individual behavioral methods over a 12-week period will be effective in reducing dental plaque. Each child will be given reward of his own choice from gift box at follow up. The record noted at follow up will be used for evaluation of intervention implemented. Since the clinician is involved in provision and dealing of community health services to special children e.g. of autism, therefore it will be easier for the clinician to build up a rapport with the patients.

OUTCOME The expected outcome of the study will be Assessment and comparison of changes observed in oral health with respect to application of PECS intervention in ASD children.

OUTCOMEMEASURE:

The outcome measures will be evaluated in follow up examination after a period of three months by defining changes observed in PI and GI scores calculated before and after intervention applied.

VARIABLES:

INDEPENDENT VARIABLES:

Demographic: Age, gender, child assessment criteria, parent's education, family income.

DEPENDENT VARIABLE:

Outcome of intervention i.e., evaluation of oral hygiene (GI and PI)

ELIGIBILITY:
Inclusion Criteria:

* Children with Confirmed diagnosis of ASD classified on the basis of CARS score 30-36.5 who understand visual or simple verbal instructions.
* Age range between 4 to 6 years
* Cooperative for oral examination

Exclusion Criteria:

* ASD children with any systemic disease which can affect oral health.
* Identification of any oral condition requiring immediate dental treatment.
* Multiple disabilities, down syndrome, epilepsy patients.
* Taking drugs such as anticonvulsant, antidepressants, anti-anxiety which can affect oral cavity tissues.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Plaque Index (PI) | Three Month
  The outcome measure will be evaluated in follow up examination after a period of three months by defining changes observed in PI scores calculated before and after intervention applied.
Gingival Index (GI) | Three month
  The outcome measures will be evaluated in follow up examination after a period of three months by defining changes observed in GI scores calculated before and after intervention applied.

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan